CLINICAL TRIAL: NCT04866342
Title: SCO2T Study: A Randomised Crossover Study Comparing Pulse Oximeter Technology Using Automatic Oxygen Control for Preterm Infants
Brief Title: Servo Controlled Oxygen Targeting (SCO2T) Study: Masimo vs. Nellcor
Acronym: SCO2T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AC20114
Record Dates: First submitted 2021-01-06; First posted 2021-04-29 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: Premature; Premature Infant; Oxygen Therapy; Hypoxia; Hyperoxia; Obstetric Labor, Premature
Keywords: Servo Control; Closed-Loop Automated Oxygen Control; Pulse oximeter technology
MeSH Terms: conditions — Premature Birth; Hypoxia; Hyperoxia; Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single centre, randomised crossover trial of two different internal oximeter monitoring systems in an automated (servo) control device - IntellO2 (Vapotherm, USA) - delivering nasal high flow employing automated oxygen titration. Each infant will act as their own control.
Masking Description: commence on either Masimo oximetry or Nellcor oximetry using the Oxygen Assist Module (OAM), IntellO2 Vapotherm device. SpO2 (range 90-95%) will be continuously monitored on a second pulse oximetry probe connected to a bedside multiparameter monitor as per normal standard of care.
  To remove selection bias the 20 infants will be randomised using sealed, windowless, envelopes. Half will instruct to commence on automated control (Precision Flow technology IntellO2, Vapotherm, USA) using Masimo oximetry technology to target SpO2 to 90-95%. Half will have instructions to commence on automated control (Precision Flow technology IntellO2, Vapotherm, USA) using Nellcor oximetry technology to target SpO2 to 90-95%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Servo control - Masimo oximetry technology (Oxygen Assist Module, IntellO2, Vapotherm) (Experimental): Automated control of oxygen. The oxygen saturation target range will be set to 90-95% (set to maintain an integral value of 93%) as per standard clinical practice.
  Automated oxygen control can be overridden by manual adjustment of oxygen at any time if this is considered necessary to optimise control of oxygenation according to current clinical targets.
  Interventions: Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - IntellO2 OAM
- Servo control - Nellcor oximetry technology (Oxygen Assist Module, IntellO2, Vapotherm) (Active Comparator): Automated control of oxygen. The oxygen saturation target range will be set to 90-95% (set to maintain an integral value of 93%) as per standard clinical practice.
  Automated oxygen control can be overridden by manual adjustment of oxygen at any time if this is considered necessary to optimise control of oxygenation according to current clinical targets.
  Interventions: Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - IntellO2 OAM

INTERVENTIONS:
Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - IntellO2 OAM — FiO2 adjustments will be made by the IntellO2 Oxygen Assist Module (OAM) for Precision Flow (IntellO2, Vapotherm, USA). By means of a modified closed-loop algorithm, the devise uses MasimoSET or Nellcor pulse oximetry to target a user-set SpO2 value.
  Manual adjustments of the inspired oxygen fraction can additionally be made as per standard care.

SUMMARY:
Most premature babies require oxygen therapy. There is uncertainty about what oxygen levels are the best. The oxygen levels in the blood are measured using a monitor called a saturation monitor and the oxygen the baby breathes is adjusted to keep the level in a target range. Although there is evidence that lower oxygen levels maybe harmful, it is not known how high they need to be for maximum benefit. Very high levels are also harmful. Saturation monitors are not very good for checking for high oxygen levels. For this a different kind of monitor, called a transcutaneous monitor, is better.

Keeping oxygen levels stable is usually done by nurses adjusting the oxygen levels by hand (manual control). There is also equipment available that can do this automatically (servo control). It is not known which is best.

Research suggests that different automated devices control oxygen effectively as measured by the readings from their internal oxygen saturation monitoring systems. When compared to free-standing saturation monitors there appears to be variations in measured oxygen levels between devices. This could have important clinical implications.

This study aims to show the different achieved oxygen levels when babies are targeted to a set target range. Babies in the study will have both a saturation monitor and a transcutaneous oxygen monitor at the same time. Both types of monitor have been in long term use in neonatal units.

For a period of 12 hours, each baby will have their oxygen adjusted automatically using two different internal oxygen monitoring technologies (6 hours respectively). The investigators will compare the range of oxygen levels that are seen between the two oxygen saturation monitoring technologies.

The investigators will study babies born at less than 30 weeks gestation, who are at least 2 days old, on nasal high flow and still require added oxygen.

DETAILED DESCRIPTION:
Presently oxygen is titrated against saturation (SpO2) by manual adjustment. Automated or servo-control systems have been developed that result in tighter control of SpO2 and more time spent in the intended target range. These systems are already in clinical use. Automated systems produce quite large fluctuations in fraction of inspired oxygen (FiO2) in order to keep SpO2 in range. It is possible that this could result in short periods of high or low oxygen tension (PO2) that are undetectable using saturation monitoring. Studies to date have examined the effects of manual and automated (servo) oxygen targeting on SpO2 but not on transcutaneous oxygen tension (TcPO2).

Research suggests that individual servo control devices control oxygen effectively as measured by the readings obtained from their internal SpO2 monitoring system. The device the investigators intend to study is available with two different oximeter monitoring systems. When compared to a separate free-standing SpO2 monitor the devices have a systematic bias in the clinically targeted range. Consequently, this could allow variations between infants in oxygenation large enough to influence important clinical outcome to go unrecognised.

There is a need to determine the achieved SpO2 and TcPO2 distributions associated with the use of different automated control systems as a first step in planning future trials. When this is measured over a small number of hours it is not anticipated that this would have an influence on clinical outcome.

This study is a prospective, single centre, randomised crossover trial of two different internal oximeter monitoring systems in an automated (servo) control device - IntellO2 (Vapotherm, USA) - delivering nasal high flow employing automated oxygen titration. Each infant will act as their own control. Infants born at less than 30 weeks gestation, greater than 48 hour of age and receiving supplementary oxygen will be eligible for inclusion.

The study will be undertaken in the Neonatal Unit at the Simpson Centre for Reproductive Health at the Royal Infirmary of Edinburgh.

Total study time is 12 hours for each infant. Infants will be randomised to commence on either Masimo oximetry or Nellcor oximetry using the Oxygen Assist Module (OAM), IntellO2 Vapotherm device. SpO2 (range 90-95%) will be continuously monitored on a second pulse oximetry probe connected to a bedside multiparameter monitor as per normal standard of care.

Additional monitoring will be carried out as shown below:

1. TcPO2 monitoring
2. FiO2 monitoring
3. Heart rate monitoring (used to validate SpO2 readings)
4. Arterial gas sampling (only if conducted by the direct care team as part of the routine care of the infant; no extra blood samples will be taken as part of the study)

FiO2 will be adjusted by the respiratory support device which has integrated automated oxygen control, set to maintain a SpO2 target range of 90-95%.The IntellO2 device uses Precision Flow technology (IntellO2, Vapotherm, USA). By means of a modified closed-loop algorithm, the devise uses MasimoSET or Nellcor pulse oximetry to target a user-set SpO2 value.

SpO2 readings will be downloaded directly from the multiparameter patient monitor. SpO2 will be measured using a Phillips MX500 multiparameter monitor (Phillips, Germany, CE 0366).TcPO2 will be measured using a SenTec Digital Monitoring System with OxiVent sensor (SenTec AG, Switzerland, European patent No. 1535055, CE 0120). Both monitors are routinely used in clinical practice. Transcutaneous data will be recorded contemporaneously and the site of the transcutaneous probe will be rotated on each infant every 2 hours. Control of sensor temperature and application duration are designed to meet all applicable standards and this monitoring device is used routinely in many neonatal units.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at less than 30 weeks gestation
2. Infants greater than 48 hours of age
3. Infants who are receiving supplementary oxygen
4. Person with parental responsibility able to give consent

Exclusion Criteria:

1. Congenital anomalies that would prevent targeting SpO2 to 90-95% (e.g. cardiac defects)
2. Clinical condition of an infant would impair accurateTcPO2 measurement (e.g. impaired perfusion or requirement of inotropic or vasopressor support)
3. Parent/person with parental responsibility unable to give informed consent on behalf of the infant
4. Infants born less than 22 weeks gestation

Min Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperoxia and hypoxia on saturation monitoring | 12 hours
  To discover the percentage time spent within target SpO2 range of 90-95% when infants are targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).

SECONDARY OUTCOMES:
Transcutaneous oxygen variability | 12 hours
  To discover the percentage time spent within a TcPO2 range of 50mmHg (6.7kPa) - 80mmHg (10.7kPa) when infants are targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Saturation variability | 12 hours
  To discover the variability in SpO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Fraction of inspired oxygen variability | 12 hours
  To discover the variability in FiO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Pooled frequency histogram of TcPO2 | 12 hours
  To generate a pooled frequency histogram of percentage time at a TcPO2 of below 30mmHg, 30-39.9mmHg, 40-49.9mmHg, 50-59.9mmHg, 60-69.9mmHg, 70-79.9mmHg, and 80mmHg and above for infants targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Pooled frequency histogram of SpO2 | 12 hours
  To generate a pooled frequency histogram of percentage time at each SpO2 point between 80 - 100% for infants targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Pooled frequency histogram of FiO2 | 12 hours
  To generate a pooled frequency histogram of the cumulative frequency at a FiO2 of 0.21-0.3, 0.31-0.4, 0.41-0.5, 0.51-0.6, 0.61-0.7, 0.81-0.9 and 0.91-1.0 for infants targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Desaturations | 12 hours
  To discover the frequency of desaturations for infants targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Desaturations | 12 hours
  To discover the duration of desaturations for infants targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).
Desaturations | 12 hours
  To discover the depth of desaturations and the area (change in PO2 versus time) above and below the set PO2 threshold for infants targeted to an SpO2 range of 90-95% with an automated (servo) control device using two internal oximeter monitoring systems (Masimo and Nellcor).

CONTACTS AND LOCATIONS:
Locations (1):
- The Simpson Centre for Reproductive Health, Royal Infirmary Edinburgh, Edinburgh, City Of Edinburgh, United Kingdom